CLINICAL TRIAL: NCT01094938
Title: Cardiac Output Monitoring in Aortic Aneurysm Surgery
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Dr Tina Mclelland, NHS Lothian
Other Study IDs: EDICOAAS; 07/S1102/30 (Other: NHS Lothian)
Record Dates: First submitted 2010-03-26; First posted 2010-03-29 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2010-03

CONDITIONS: Aneurysm
Keywords: Aortic aneurysm repair
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Repair

SUMMARY:
To compare CO values obtained by the lithium indicator dilution method and pulse power analysis before, during and after anaesthesia and surgery for the elective repair of abdominal aortic aneurysms. This will enable us to determine how often and when calibration of the pulse power analysis derived CO is required.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for elective abdominal aortic and extent 4 thoracoabdominal aortic aneurysm repair

Exclusion Criteria:

* Patients not giving informed consent.
* Patients under the age of 18 years.
* Patients who may be pregnant
* Patients with learning disabilities.
* Rhythm other than sinus rhythm.
* Patients on oral lithium therapy.
* Patients less than 40kg
* Patients with severe mitral regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Edinburgh based trial in aortic aneurysm repair
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-07; Primary Completion 2007-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Cardiac output

SECONDARY OUTCOMES:
Arterial Pressure

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom